CLINICAL TRIAL: NCT04066829
Title: Default Dosing Settings for Opioid Prescriptions to Adolescents and Young Adults After Tonsillectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Kao-Ping Chua, Assistant Professor of Pediatrics, University of Michigan
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HUM00159821; 1K08DA048110 (NIH)
Record Dates: First submitted 2019-08-22; First posted 2019-08-26 (Actual); Results first posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Tonsillectomy
Keywords: Default settings; Opioid prescribing; Electronic Health Record; Opioid; Opioid Use; Behavioral intervention

STUDY DESIGN:
Masking Description: Intervention is assigned based on location. Participants and providers are 'nudged' but not masked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Default setting intervention (Experimental): The arm will include all patients undergoing tonsillectomy at C.S. Mott Hospital by a pediatric otolaryngology faculty member at the University of Michigan.
  Interventions: Behavioral: Default setting intervention
- No Intervention: Control (Usual Care) (No Intervention): The arm will include all patients undergoing tonsillectomy at University Hospital, Brighton Center for Specialty Care, or Livonia Center for Specialty Care by a general otolaryngology faculty member at the University of Michigan.

INTERVENTIONS:
Behavioral: Default setting intervention — The new default settings will be implemented only for patients in the experimental arm.
  Arms: Experimental: Default setting intervention

SUMMARY:
This study will evaluate whether lowering the default number of doses for opioid prescriptions written in an electronic health record system can decrease opioid prescribing without causing unintended consequences such as worsened pain control.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents and young adults aged 12-25 years undergoing tonsillectomy at C.S. Mott Hospital, University Hospital, Brighton Center for Specialty Care, or Livonia Center for Specialty Care from October 2019-July 2021, excluding April-May 2020 (owing to suspension of elective procedures due to COVID-19).
* Surgeon belongs to the Department of Otolaryngology at the University of Michigan Medical School
* Patients are not any of the following: patients living in foster care or with a legal guardian, patients with medical complexity or developmental delays, non-English speaking patients, patients with recent suicidal ideation documented in their chart, or patients undergoing emergent tonsillectomy.

Exclusion Criteria:

* Patients with prescription opioid use prior to surgery
* Patients undergoing additional procedures at the same time as tonsillectomy (other than minor procedures such as tympanostomy tube placement)
* Patients enrolled in another study
* Patients who are not prescribed opioids post-operatively at discharge
* Patients who are enrolled in the Michigan Pain-control Optimization Pathway (M-POP), which includes education about pain management and a small initial opioid prescription
* Patients with hospitalization with length of stay > 1 day after surgery
* Patients who decline to enroll
* Additional exclusion criteria for secondary analysis: Patients who do not complete the baseline and post-operative day 14 surveys

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 198 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kao-Ping Chua, Principal Investigator — University of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chua KP, Thorne MC, Ng S, Donahue M, Brummett CM. Association Between Default Number of Opioid Doses in Electronic Health Record Systems and Opioid Prescribing to Adolescents and Young Adults Undergoing Tonsillectomy. JAMA Netw Open. 2022 Jun 1;5(6):e2219701. doi: 10.1001/jamanetworkopen.2022.19701. PMID 35771572

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 282 participants were eligible of whom data from 237 participants was used. 198 consented; the other 39 could not be approached for consent.
  The IRB approved analysis of Electronic Medical Record data for these patients for the primary outcomes only, determining that review of electronic medical record data was no more than minimal risk and was justified to maximize sample size and power in light of decreased tonsillectomy volume at the University of Michigan owing to COVID-19.
Pre-assignment Details: 45 participants who were initially eligible to participate in the study were excluded because they declined to participate, withdrew or did not undergo a tonsillectomy, did not receive a discharge opioid prescription, had prior opioid use, or opted for an opioid sparing pathway.
Groups:
- Pediatric Otolaryngology Service (Pre-Intervention): October 1, 2019 - September 30, 2020 The arm included all patients undergoing tonsillectomy at C.S. Mott Hospital by a pediatric otolaryngology faculty member at the University of Michigan.
- Pediatric Otolaryngology Service (Post-Intervention): October 1, 2020 - July 31, 2021 The arm included all patients undergoing tonsillectomy at C.S. Mott Hospital by a pediatric otolaryngology faculty member at the University of Michigan.
- General Otolaryngology Service (Control, Pre-Intervention): October 1, 2019 - September 30, 2020 The arm included all patients undergoing tonsillectomy at University Hospital, Brighton Center for Specialty Care, or Livonia Center for Specialty Care by a general otolaryngology faculty member at the University of Michigan.
- General Otolaryngology Service (Control, Post-Intervention): October 1, 2020 - July 31, 2021 The arm included all patients undergoing tonsillectomy at University Hospital, Brighton Center for Specialty Care, or Livonia Center for Specialty Care by a general otolaryngology faculty member at the University of Michigan.
Period: Overall Study
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Started | 70 | 61 | 46 | 60
Participants Who Completed the Post-operative Day 14 Survey Assessing Secondary Outcomes. | 44 | 40 | 26 | 40
Completed | 70 | 61 | 46 | 60
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention) | Total
Number analyzed (Participants) | 70 | 61 | 46 | 60 | 237
Age, Customized [Count of Participants; unit: Participants]
  Ages 12 years to 17 years | 62 | 57 | 3 | 5 | 127
  Ages 18 years to 25 years | 8 | 4 | 43 | 55 | 110
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 28 | 27 | 16 | 16 | 87
  Female | 40 | 34 | 30 | 43 | 147
  Other | 2 | 0 | 0 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White/Non-Hispanic | 54 | 44 | 37 | 46 | 181
  Black/Non-Hispanic | 5 | 7 | 2 | 7 | 21
  Hispanic/Any Race | 3 | 6 | 3 | 3 | 15
  Asian/Non-Hispanic | 4 | 0 | 2 | 1 | 7
  Other/Multi-Racial/Non-Hispanic | 3 | 1 | 1 | 2 | 7
  Unknown Race or Ethnicity | 1 | 3 | 1 | 1 | 6
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70 | 61 | 46 | 60 | 237

OUTCOME MEASURES:

1. Primary Outcome: Number of Doses in the Initial Discharge Opioid Prescription
Description: Doses are defined as the maximum number of instances a patient could take opioids if they took them as prescribed. Number of doses are calculated from the electronic health record.
Time Frame: Day of discharge, approximately 1 day
Measure: Mean (Standard Deviation); unit: Doses
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 70 | 61 | 46 | 60
Doses | 22.3 (7.4) | 16.1 (6.5) | 33.7 (20.4) | 30.4 (12.4)
Statistical Analysis 1: Comparison: Pediatric Otolaryngology Service (Pre-Intervention) vs Pediatric Otolaryngology Service (Post-Intervention) vs General Otolaryngology Service (Control, Pre-Intervention) vs General Otolaryngology Service (Control, Post-Intervention); Pre and post difference in the treatment group as compared to the control group. A log transformation was used; Test type: Other; Difference in Differences = -29.2, 95% CI 2-sided [-42.2 to -11.8]

2. Primary Outcome: Proportion of Patients for Whom the Number of Doses in the Discharge Opioid Prescription Equals the Number of Doses in the New Default Settings
Description: The new default settings called for 12 doses in the discharge prescription.
  This measure assesses the proportion of participants with 12 doses in the discharge prescription, regardless of which arm they were in.
  Doses are defined as the maximum number of instances a patient could take opioids if they took them as prescribed. Number of doses are calculated from the electronic health record.
Time Frame: Day of discharge, approximately 1 day
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 70 | 61 | 46 | 60
Participants | 1 | 27 | 2 | 0

3. Primary Outcome: Proportion of Participants Who Had at Least One Opioid Prescription Refill From University of Michigan During the Two Weeks After Surgery
Description: as for outcome 1
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 70 | 61 | 46 | 60
Participants | 10 | 12 | 25 | 26

4. Primary Outcome: Proportion of Patients Who Visited or Saw a University of Michigan Provider Due to Pain During the Two Weeks After Surgery
Description: Detailed in electronic health record. Excludes emergency department visits and hospitalizations for pain.
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 70 | 61 | 46 | 60
Participants | 2 | 1 | 0 | 1

5. Primary Outcome: Proportion of Patients With at Least One Emergency Department and/or Hospitalization at University of Michigan for Pain During the Two Weeks After Surgery
Description: Detailed in electronic health record
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 70 | 61 | 46 | 60
Participants | 3 | 2 | 2 | 3

6. Secondary Outcome: Overall Satisfaction Score on Pain Control During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Description: Participants were surveyed on Day 14 and asked to report level of satisfaction with pain control since their surgery.
  Pain control satisfaction is on a scale of 1-10 with higher scores indicating higher satisfaction
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 26 | 40
units on a scale | 7.4 (2.4) | 7.4 (2.4) | 6.5 (2.5) | 6.7 (7.0)

7. Secondary Outcome: Proportion of Patients Who Reported That Their Pain Was Well-controlled as Measured by the Post-operative Survey.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 25 | 40
Participants | 32 | 25 | 11 | 18

8. Secondary Outcome: Proportion of Patients Whose Overall Pain Control Was Rated as Much Worse or Worse Than Expected as Measured by the Post-operative Survey.
Description: Survey was comprised of 5 options:
  * Much worse than you expected
  * Worse than you expected
  * About what you expected
  * Better than you expected
  * Much better than you expected
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 39 | 26 | 40
Participants | 15 | 11 | 11 | 18

9. Secondary Outcome: Proportion of Patients Whose Pain Has Resolved by Day 14 After Surgery as Measured by the Post-operative Survey.
Description: Survey asked participant on what day pain had resolved. If participants indicated pain had resolved by Day 14, then they were coded as 1, and 0 otherwise.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 26 | 40
Participants | 32 | 34 | 17 | 24

10. Secondary Outcome: Pain in the Throat and/or Mouth Over the Past 7 Days at Its Worst as Measured by the Post-operative Survey.
Description: Pain control is on a scale of 0-10 with higher scores indicating more pain.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 26 | 40
score on a scale | 5.3 (2.8) | 5.4 (3.2) | 7.1 (2.0) | 6.4 (3.1)

11. Secondary Outcome: Pain in the Throat and/or Mouth Over the Past 7 Days on Average as Measured by the Post-operative Survey.
Description: Pain control is on a scale of 0-10 with higher scores indicating worse pain.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 26 | 40
score on a scale | 3.3 (2.1) | 3.3 (3.0) | 4.4 (2.0) | 3.9 (2.2)

12. Secondary Outcome: Proportion of Patients With Leftover Doses of Opioids as Measured by the Post-operative Survey.
Description: Participants who answered 'No' to the following question: Did you take all of the opioid pain medications that were prescribed to you during the two weeks after surgery?
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 38 | 26 | 38
Participants | 35 | 28 | 21 | 24

13. Secondary Outcome: Number of Opioid Doses Taken During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Description: Patients were asked to report the number of instances in which they used opioids prescribed to them.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: Opioid Doses Consumed
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 41 | 36 | 25 | 33
Opioid Doses Consumed | 7.2 (8.0) | 9.5 (9.6) | 27.3 (18.7) | 23.3 (23.4)

14. Secondary Outcome: Proportion of Patients Who Misused Opioids Prescribed to Others at Least Once During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Description: Includes any use of opioids prescribed to others
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 38 | 26 | 39
Participants | 0 | 0 | 0 | 0

15. Secondary Outcome: Proportion of Patients Who Misused Opioids Prescribed to Them at Least Once During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Description: Includes taking one's own opioids in greater amounts, more often, or longer than directed by a doctor.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 38 | 26 | 39
Participants | 0 | 0 | 0 | 0

16. Secondary Outcome: Patient Health Questionnaire 8-item (PHQ-8) Score (Depression) as Measured by the Post-operative Survey.
Description: This is an 8-item self-report scale, all items are rated on a score of 0-3, for a total range of 0-24. Higher scores indicate more depressive symptoms
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 43 | 39 | 26 | 40
score on a scale | 5.1 (5.6) | 5.6 (4.9) | 7.4 (4.4) | 7.6 (5.1)

17. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)- Pediatric Anxiety - Short Form 8a Score as Measured by the Post-operative Survey.
Description: This measure is 8 items each scored from 1 to 5 points, with the lowest possible raw score being 8 and the highest possible raw score being 40. Higher scores indicate greater anxiety,
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 42 | 39 | 25 | 40
score on a scale | 11.2 (4.6) | 12.4 (6.1) | 15.9 (8.1) | 13.4 (7.2)

18. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS)- Sleep Disturbance - Short Form 4a Score as Measured by the Post-operative Survey.
Description: This measure is 4 items each scored from 1 to 5 points, with the lowest possible raw score being 8 and the highest possible raw score being 40. Higher scores indicate greater sleep disturbance, i.e. worse sleep.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 42 | 39 | 25 | 40
score on a scale | 8.4 (2.9) | 9.7 (3.7) | 12.2 (4.0) | 11.2 (42)

19. Secondary Outcome: Proportion of Patients Who Saw Their Primary Care Doctor (or a Colleague) in the Office Due to Pain at Least Once During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 25 | 40
Participants | 3 | 0 | 1 | 0

20. Secondary Outcome: Proportion of Patients Who Visited a Retail Clinic Due to Pain at Least Once During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 25 | 40
Participants | 1 | 1 | 0 | 1

21. Secondary Outcome: Proportion of Patients Who Visited an Urgent Care Center Due to Pain at Least Once During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 25 | 40
Participants | 1 | 0 | 3 | 0

22. Secondary Outcome: Proportion of Patients Who Visited an Emergency Department and/or Were Hospitalized Due to Poorly Controlled Pain at Least Once During the Two Weeks After Surgery as Measured by the Post-operative Survey.
Time Frame: Day 14
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 44 | 40 | 25 | 40
Participants | 3 | 0 | 4 | 3

23. Secondary Outcome: Proportion of Patients With Leftover Doses Who Disposed of Them
Description: Proportion of patients with leftover doses who disposed of them
Time Frame: 14 Days
Population: The numbers above reflect the number of participants with complete data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
Number analyzed (Participants) | 34 | 25 | 19 | 23
Participants | 28 | 17 | 13 | 17

ADVERSE EVENTS:
Time Frame: 14 Days
Arm/Group | Pediatric Otolaryngology Service (Pre-Intervention) | Pediatric Otolaryngology Service (Post-Intervention) | General Otolaryngology Service (Control, Pre-Intervention) | General Otolaryngology Service (Control, Post-Intervention)
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/61 | 0/46 | 0/60
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/61 | 0/46 | 0/60
Other Adverse Events (participants affected / at risk) | 0/70 | 0/61 | 0/46 | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT04066829/Prot_SAP_001.pdf
  • Informed Consent Form (2020-12-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT04066829/ICF_002.pdf